CLINICAL TRIAL: NCT02920853
Title: Testing the Efficacy of Enhanced Biofeedback on Chronic Musculoskeletal Pain
Brief Title: Enhanced Biofeedback for Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tulsa (Other)
Responsible Party: Principal Investigator, Jamie Rhudy, Professor, University of Tulsa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TU1645
Record Dates: First submitted 2016-09-26; First posted 2016-09-30 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Musculoskeletal Pain
Keywords: chronic pain
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BT-CPR (Experimental): Participants will receive training in relaxation and biofeedback to develop skills in relaxation/arousal reduction, and pain reduction. Then they will practice relaxing and reducing their arousal as they view graphical arousal feedback. Electric stimulations will be delivered throughout the biofeedback training to provide pain relief when relaxation is achieved.
  Interventions: Behavioral: Biofeedback Training (BT-CPR)
- Biofeedback-Only (Active Comparator): Participants will receive training in relaxation and biofeedback to develop skills in relaxation/arousal reduction, and pain reduction. Then they will practice relaxing and reducing their arousal as they view graphical arousal feedback.
  Interventions: Behavioral: Biofeedback Training

INTERVENTIONS:
Behavioral: Biofeedback Training (BT-CPR) — Participants will receive biofeedback training (which will include electric stimulations) to reduce arousal and pain
  Arms: BT-CPR
Behavioral: Biofeedback Training — Participants will receive biofeedback training to reduce arousal and pain
  Arms: Biofeedback-Only

SUMMARY:
The purpose of this study is to assess whether a novel, enhanced form of biofeedback can help individuals regulate their chronic musculoskeletal pain more effectively.

DETAILED DESCRIPTION:
Relaxation is a low-cost treatment for managing pain with little or no side effects. The proposed study will use a novel biofeedback treatment to try and enhance the capacity of relaxation to engage pain inhibitory circuits. Specifically, a biofeedback system (Biofeedback Training for Conditioned Pain Regulation, BT-CPR) will be used to monitor the participant's level of sympathetic arousal and will use this to control the intensity of painful stimulations delivered to the participant during biofeedback training. Thus, when the participant successfully relaxes (and reduces their arousal), the intensity is lowered and produces pain relief. Efficacy of the treatment will be tested in a small, randomized controlled trial in which individuals with a verified diagnosis of chronic musculoskeletal pain will receive 10 treatment sessions, or 10 sessions of a control condition (traditional biofeedback, to control for the effects of relaxation on pain). The aim will be to assess whether the treatment results in improvements in clinical pain outcomes (e.g., pain intensity, quality of life, pain interference) and psychosocial variables (e.g., coping, self-efficacy, mood).

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older) with a verified diagnosis of chronic musculoskeletal pain and currently experiencing pain

Exclusion Criteria:

* under 18 years of age (given the nature of the treatment study)
* if female, currently pregnant
* persistent feelings of numbness in hands and feet
* difficulty being able to feel or sense things
* lack of access to a computer or smartphone (to complete electronic pain diaries)
* injuries that prevent sensor application
* use of narcotic pain medications with 48 hours of treatment sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Changes in clinical pain | Assessed daily via electronic diaries starting 1 week prior to session 1 and ending 1 week after session 10 (up to 11 weeks)
  Self-report ratings of pain intensity, rated using 0-10 Likert-type scales, (i.e., 0 = no pain; 10 = most intense pain).
Changes in psychosocial outcomes | Assessed daily via electronic diaries starting 1 week prior to session 1 and ending 1 week after session 10 (up to 11 weeks)
  Self-report ratings of pain interference, mood, sleep quality, and coping. These items are rated using 0-10 Likert-type scales, (e.g., 0 = no change; 10 = extreme change) with higher values indicating an increase in the variable assessed on a particular item (e.g., interference with daily activities).

SECONDARY OUTCOMES:
Changes in reactions to painful stimuli | Assessed immediately before the first treatment session (Time 1) and immediately after (Time 2) the last treatment session (approximately 10 weeks from Time 1).
  Subjective ratings of painful stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Rhudy, PhD, Principal Investigator — The University of Tulsa
Locations (1):
- University of Tulsa, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No